CLINICAL TRIAL: NCT03305224
Title: The Study of Combination Therapy With Radium-223 and Enzalutamide in Osaka City University
Brief Title: The Combination Therapy With Ra-223 and Enzalutamide
Acronym: CORE-OCU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taro Iguchi, MD, PHD (Other)
Collaborators: Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Taro Iguchi, MD, PHD, Principal Investigator, Osaka City University
Organization: Osaka City University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORE-OCU
Record Dates: First submitted 2017-08-28; First posted 2017-10-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Castration-resistant Prostate Cancer; Bone Metastases
Keywords: castration-resistant prostate cancer; bone metastasis
MeSH Terms: interventions — Radium-223; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ra-223 + Enzalutamide (Other)
  Interventions: Drug: Ra-223 in combination with enzalutamide

INTERVENTIONS:
Drug: Ra-223 in combination with enzalutamide — Ra-223 (55 kBq/kg i.v.) 6 injections at 4 weeks interval in combination with enzalutamide 160 mg per a day

SUMMARY:
This study is to evaluate preliminary efficacy of Ra-223 in combination with Enzalutamide in progressive CRPC patients with bone metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as CRPC
2. Surgical or those who will be treated with luteinizing hormone-releasing hormone (LHRH) agonists throughout the study period,
3. Patients who had >30% of PSA response to enzalutamide prior to enrollment,
4. Interval between PSA progression and enrollment is up to 3 months,
5. With bone metastases (≥ 2 hot spots) on bone scintigraphy within previous 24 weeks,
6. No intention to use anti-cancer chemotherapy within the next 6 months,
7. Eastern Cooperative Oncology Group performance status (ECOG-PS): 0-1,
8. Life expectancy ≥ 6 months,
9. Laboratory requirements within 30 days before enrollment:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10e9/L,
   * Platelet count ≥ 100 x 10e9/L,
   * Hemoglobin ≥ 10.0 g/dL,
   * Total bilirubin level ≤1.5 institutional upper limit of normal (ULN),
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 ULN,
   * Creatinine ≤ 1.5ULN, and estimated glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2,
10. Age ≥ 20,
11. Ability to understand and the willingness to sign a written informed consent (IC).

Exclusion Criteria:

1. Prior chemotherapy or planned treatment with chemotherapy,
2. PSA progression within 3 months after initiation of enzalutamide
3. Prior treatment with corticosteroids, estramustine or abiraterone acetate,
4. Any systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bone metastases,
5. Had history of gastrointestinal bleeding or ulcer within 3 months prior to study entry,
6. History of visceral metastasis, or presence of visceral metastasis detected by screening imaging examinations,
7. History of or known brain metastasis,
8. Malignant lymphadenopathy ≧1.5 cm in short axis,
9. Imminent or established spinal cord compression based on clinical findings and/or MRI (Magnetic Resonance Imaging),
10. Any other serious illness or medical condition
11. Substance abuse, medical, psychological, or social conditions that might interfere with the subject's participation in the study or evaluation of the study Results
12. Those who judged to be inappropriate by the principal investigator or co-investigator.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Alkaline phosphatase (ALP) | 6 months
  Percentage of change from baseline to 6 months (or earlier for those who discontinue study therapy)

SECONDARY OUTCOMES:
Tolerability of Radium-223 therapy | 6 months
  Proportion of patients who complete 6 times injections of radium-223
Evaluation for bone metastasis by 18F-NaF-PET | 1, 3, 6 months
  Fractional decline of intensity of tracer uptake measured by SUVmax on 18F-NaF-PET at 1, 3, 6 months.
Evaluation for bone metastasis by bone scintigraphy | 1, 3, 6 months
  The change of Bone Scan Index (BSI) by bone scintigraphy at 1, 3, 6 months.
Overall Survival Rate | 3 years
  Overall Survival (OS) is defined as the time from the registration to death due to any cause, or censored at date last known alive.
Time to occurrence of Symptomatic Skeletal-related Events (SSEs) | 1 year
  Time to occurrence of SSEs are defined asthe time from registration to the date of the occurrence of SSEs (symptomatic fracture, surgery or radiation to bone, or spinal cord compression).
Time to occurrence of visceral metastasis | 1 year
  Time to occurrence of visceral metastasis was defined as the time from registration to the date of the occurrence of a visceral metastasis for each patient.
Time to initiation of cytotoxic chemotherapy | 1 year
  The time to initiation of cytotoxic chemotherapy is defined as the time from registration to the date of initiation of cytotoxic chemotherapy.
Changes in Prostate Specific Antigen (PSA) | 6 months
  Percent change in prostate-specific antigen (PSA) from baseline at 6 months.
Changes From Baseline for Brief Pain Inventory (BPI) | 6 months
  The change for the BPI-SF (Brief Pain Inventory-Short Form) score was calculated.
Changes From Baseline for Functional Assessment of Cancer Therapy - Prostate (FACT-P) | 6 months
  The change for the FACT-P TOI domain (physical and social well-being and prostate specific score) was calculated.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 6 months
  Number of participants with adverse events as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka City University Graduate School of Medicine, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No